CLINICAL TRIAL: NCT04046029
Title: Bivalirudin vs Heparin in Elderly Patients With Acute Coronary Syndrome Undergoing Elective Percutaneous Coronary Intervention
Brief Title: Bivalirudin in Elderly Patients Undergoing Elective Percutaneous Coronary Intervention.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PJ-KS-KY-2019-38(X)
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Acute Coronary Syndrome; Percutaneous Coronary Intervention; Aging; Anticoagulants and Bleeding Disorders
Keywords: Acute Coronary Syndrome; Percutaneous Coronary Intervention; Elderly; Bivalirudin
MeSH Terms: conditions — Acute Coronary Syndrome; Hemostatic Disorders | interventions — bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bivalirudin (Experimental)
  Interventions: Drug: Bivalirudin
- Heparin (Active Comparator)
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Bivalirudin — Bivalirudin will be given as a bolus of 0.75 mg/kg followed by infusion of 1.75 mg/kg/h during the PCI procedure and for at least 30 minutes but no more than 4 hours afterwards. Following this mandatory infusion,a reduced-dose infusion (0.2 mg/kg/h) for up to 20 hours could be administered at physician discretion. An additional bivalirudin bolus of 0.3 mg/kg was given if the activated clotting time 5 minutes after the initial bolus was less than 225 seconds.
  Arms: Bivalirudin
Drug: Heparin — Heparin will be administered at a dose of 70 to 100 units per kilogram in patients not receiving glycoprotein IIb/IIIa inhibitors and at a dose of 50 to 70 units per kilogram in patients receiving glycoprotein IIb/IIIa inhibitors. Subsequent adjustment of the heparin dose on the basis of the activated clotting time will be left to the discretion of the treating physicians.
  Arms: Heparin

SUMMARY:
The study is an investigator-sponsored, prospective, multicenter, randomized, open-label study designed to compare efficacy and safety between bivalirudin and heparin in elderly patients with acute coronary syndrome undergoing elective percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥75 years old;
* Planned elective PCI for patients with acute coronary syndrome;
* Life expectancy ≥ 1 year;
* Provide written informed consent.

Exclusion Criteria:

* Contraindications to angiography or PCI;
* Active bleeding or bleeding constitution, bleeding tendency, including GI or urinary tract hemorrhage (3 months), cerebral hemorrhage (6 months) or cerebral infarction history (3 months), etc;
* Other disease may lead to vascular lesions and secondary bleeding factors (such as active gastric ulcer, active ulcerative colitis, intra-cerebral mass, aneurysm, etc.);
* Severe renal insufficiency (eGFR < 30 mL/min/ 1.73 m2);
* Elevated AST, ALT level higher than three times of the normal upper limit;
* Advanced heart failure (NYHA classification grading of cardiac function ≥Ⅲ) Complicated with immune system diseases#
* Abnormal hematopoietic system: platelet count < 100 × 109 / L or >700 × 109 / L, white blood cell count < 3×109/L etc;
* Suffering from acute infections ,infectious diseases or other serious diseases, such as malignant tumors;
* Known intolerance, or contraindication to any antithrombotic medication
* Known allergy to the study drugs and instruments (UFH, bivalirudin, aspirin and clopidogrel, stainless steel, contrast agents, etc.), or those allergic constitution.
* Non-cardiac co-morbid conditions are present that may result in protocol non-compliance;
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period;
* Patient's inability to fully cooperate with the study protocol

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 7 days
  A composite of cardiac death, reinfarction, heart failure,ischemic stroke,frequent post infarction angina, Ventricular tachycardia or fibrillation requiring electrical cardioversion or defibrillation.
Major bleeding | 7 days
  BARC types 3-5 bleeding;TIMI major bleeding or GUSTO moderate to severe bleeding.

SECONDARY OUTCOMES:
Major adverse cardiac events | 30 days
  A composite of cardiac death, reinfarction, heart failure,ischemic stroke,frequent post infarction angina, Ventricular tachycardia or fibrillation requiring electrical cardioversion or defibrillation.
Stent thrombosis ,TVR ,TLR | 30 days
  Rate of stent thrombosis,unplanned target-vessel revascularization and target lesion revascularisation.
Major adverse cardiac events | 180 days
  A composite of cardiac death, reinfarction, heart failure,ischemic stroke,frequent post infarction angina, Ventricular tachycardia or fibrillation requiring electrical cardioversion or defibrillation.
Stent thrombosis ,TVR ,TLR | 180 days
  rate of stent thrombosis,unplanned target-vessel revascularization and target lesion revascularisation
Major bleeding | 30 days
  BARC types 3-5 bleeding;TIMI major bleeding or GUSTO moderate to severe bleeding.
Major bleeding | 180days
  BARC types 3-5 bleeding;TIMI major bleeding or GUSTO moderate to severe bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Shaoke Meng, M.D., Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, China

REFERENCES:
- [Background] De Caterina R, Husted S, Wallentin L, Andreotti F, Arnesen H, Bachmann F, Baigent C, Huber K, Jespersen J, Kristensen SD, Lip GY, Morais J, Rasmussen LH, Siegbahn A, Verheugt FW, Weitz JI; European Society of Cardiology Working Group on Thrombosis Task Force on Anticoagulants in Heart Disease. Parenteral anticoagulants in heart disease: current status and perspectives (Section II). Position paper of the ESC Working Group on Thrombosis-Task Force on Anticoagulants in Heart Disease. Thromb Haemost. 2013 May;109(5):769-86. doi: 10.1160/TH12-06-0403. Epub 2013 Mar 28. PMID 23636477
- [Background] Hirsh J, Anand SS, Halperin JL, Fuster V; American Heart Association. AHA Scientific Statement: Guide to anticoagulant therapy: heparin: a statement for healthcare professionals from the American Heart Association. Arterioscler Thromb Vasc Biol. 2001 Jul;21(7):E9-9. doi: 10.1161/hq0701.093520. No abstract available. PMID 11451763
- [Background] Robson R, White H, Aylward P, Frampton C. Bivalirudin pharmacokinetics and pharmacodynamics: effect of renal function, dose, and gender. Clin Pharmacol Ther. 2002 Jun;71(6):433-9. doi: 10.1067/mcp.2002.124522. PMID 12087346